CLINICAL TRIAL: NCT01357876
Title: Effect of Metformin on Gut Peptides , Bile Acids and Lipid Profiles in Type 2 Diabetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 114453
Record Dates: First submitted 2010-11-04; First posted 2011-05-23 (Estimated); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Type two diabetics (Other): Type two diabetics
  Interventions: Other: Metformin

INTERVENTIONS:
Other: Metformin — withdrawral

SUMMARY:
Metformin is a biguanide that is marketed as an oral anti-diabetic drug. Metformin treatment in concert with diet and exercise is the consensus first-line treatment for type 2 diabetes mellitus (T2DM), and therefore it will likely be an adjunct therapy for all assets in development by GSK for the treatment of T2DM. Metformin has potent effects in lowering circulating glucose concentrations, and it is believed to have additional benefits in improving macrovascular outcomes, fatty liver disease and polycystic ovarian syndrome. Its use in a significant proportion of T2DM subjects is limited by contraindications of heart failure and renal insufficiency or gastrointestinal side effects. The mechanisms underlying its glucose-lowering effect and adverse event profile of metformin are not well understood. Whilst activation of AMP kinase may be important for therapeutic effect, changes in incretin secretion and bile acid excretion have been described, but not consistently linked to its therapeutic effect or AE profile. The aim of this study is to recruit T2DM patients on prescribed metformin monotherapy to further investigate how the glucose effects are related to the alterations in bile acid absorption, incretin and lipid profiles by studying these parameters on and off the drug. This will be done in combination with frequent capillary blood glucose monitoring to ensure patient safety. This study will facilitate the development of a pharmacodynamic model that can be used by clinical teams developing non-absorbable NCEs such as iBAT inhibitors.

DETAILED DESCRIPTION:
As metformin has become first-line therapy for T2DM patients in many countries, it is important to ensure early-on in development that novel anti-diabetic NCEs work well as add-ons to this drug. Furthermore, the broad spectrum of effects of metformin that may be related to its glucose-lowering action offers the opportunity to use this drug as an investigative tool to explore the relationship between the various pharmacodynamic endpoints. In this situation, reliable PD endpoints are essential because systemic PK measurements are not available to track how a NCE target is being activated or inhibited. Therefore, a clearer understanding of metformin's mechanism of action as it relates to glycaemic control, lipid metabolism, bile acid excretion and gastrointestinal adverse effects will enable the EnteroEndocrine (EE) project teams to design more efficient studies for the evaluation of non-absorbable NCEs targeted to receptors that are accessible from the gut lumen, including the ileal bile acid transport inhibitor.

Because of the complexity of metformin kinetics within the gut, it is proposed to follow the rise and fall of fasting blood glucose during metformin washout and re-introduction, respectively, to determine the two appropriate timepoints for more detailed investigation.

As a result, subjects will be studied on 4 occasions:

1. Whilst on their usual stable dose of metformin (baseline state),
2. 7 days after stopping metformin to replicate the washout paradigm frequently used in early phase T2DM studies in GSK
3. When fasting capillary glucose has increased by 25% from the pre-metformin washout level or two weeks from the start of the wash-out period.
4. After metformin is re-introduced, when fasting capillary glucose has returned to the pre-metformin washout level (baseline state established at screening )

This study will entail the withdrawal and re-introduction of metformin under closely supervised conditions. The withdrawal of metformin will be for a maximum period up to three weeks and the glucose increases projected are not expected to result in significant long-term risk for the subjects.

If subjects do not already test blood glucose at home, a glucometer, instructions on its use, and testing strips will be provided to them for capillary blood glucose (CBG) monitoring during withdrawal and reinstatement of metformin. They will be instructed to test their blood glucose twice a day, fasting before breakfast and before dinner, and at any time they are concerned that blood glucose may have risen excessively. A written diary card will be kept by each subject for recording CBG values, beginning approximately 7 days before discontinuation of metformin after baseline assessments are completed during visit 1.

Fasting CBG values >15mM or < 3.5mM must be reported to the site at once. If fasting CBG are >15mM or < 3.5 mM on any two consecutive days during the wash-out period, the subject will be discontinued and the usual dose of metformin will be reinstated, if appropriate

Subjects are required to call the study centre while not in the unit or to alert site staff while in the clinical unit:

1. When they have CBG values that are >15mM
2. When they have CBG values that are <3.5mM
3. When they have any concerns relating to their CBG levels
4. When they have rapid, unexplained changes in their blood glucose levels

Study staff will attempt to contact the subjects daily to check on the CBG values and to record any adverse events whilst the subject is at home.

Subjects will be encouraged to keep their usual lifestyle in term of diet and exercise for all duration of the study.

The Entero-Test device is simple, safe device for the collection of duodenal bile. It is well tolerated, although some subjects may feel slight nausea on removal. Some blood may be seen on the string when removed. This occurs if the string "nicks" the oesophagus on removal, this is very minor trauma that heals rapidly and is not a cause for concern.

Primary enpoints-During metformin wash out and when treatment reinstated, pharmacodynamic endpoints will include the following as data permit:

* 24h profiles of blood glucose and insulin
* Faecal and serum bile acid profiles
* Enteroendocrine peptide profiling including but not limited to tGLP-1, tGIP, and tPYY
* Serum lipid analysis including but not limited to fasting HDL and LDL cholesterol, fasting and prandial TGs, ApoA1, ApoB and ApoE

Secondary Endpoints- • Relative bile acid composition as determined by EnteroTest bile string sampling of duodenal bile.

• Sparse metformin PK profiles will be determined from plasma samples

ELIGIBILITY:
Inclusion Criteria:

1. T2DM men and women between 18 -70 years of age on stable dose of metformin
2. Subjects taking stable regimens of aspirin, ACE inhibitors, beta-blockers, calcium channel blockers, thyroid replacement hormone, and HMG-CoA reductase inhibitors (statins) will be allowed if their dose regimen(s) remain constant throughout the study period
3. HBA1C >6.5% <8.5%
4. BMI from 22.5 up to 37.5 kg/m2, inclusive
5. AST, ALT, alkaline phosphatase and bilirubin less than or equal to 3xULN
6. Has a normal ECG as determined by unit physician.
7. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

1. medically unable or unwilling to discontinue current metformin therapy for as required by the protocol and remain off medication until the completion of Visit 3
2. past or present disease (other than T2DM) as judged by the Investigator, which may affect the outcome of this study. These diseases include, but are not limited to, cardiovascular disease, malignancy, hepatic disease, renal disease, haematological disease, neurological disease and endocrine disease.
3. subject is currently on bile acid sequestrant therapy.
4. Gastrointestinal surgery or disease that would compromise the use of the EnteroTest
5. fasting triglycerides >450mg/dL (>5.1 mmol/L)
6. Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
7. A positive pre-study drug/alcohol screen.
8. History of regular alcohol consumption within 6 months of the study defined as:

   -An average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 g of alcohol: a half-pint (~240 ml) of beer, 1 glass (125 ml) of wine or 1 (25 ml) measure of spirits.
9. Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
10. Pregnant females as determined by positive (serum or urine) hCG test at screening or prior to dosing.
11. Lactating females.
12. Unwillingness or inability to follow the procedures outlined in the protocol.

12.Subject is mentally or legally incapacitated or unable to provide informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2010-10-01 (Actual); Primary Completion 2011-07-07 (Actual); Study Completion 2011-07-07 (Actual)

PRIMARY OUTCOMES:
To investigate the relationship between the glucose lowering action of metformin and Faecal and serum bile acid concentrations | We will track this measure over a 5 week period. This may change as a patient's response to withdrawl and resumption of metformin varies
To investigate the relationship between the glucose lowering action of metformin and enteroendocrine peptide profiles including, but not limited to, incretins and PYY | We will track this measure over a 5 week period. This may change as a patient's response to withdrawl and resumption of metformin varies
To investigate the relationship between the glucose lowering action of metformin and lipid metabolism including, but not limited to, fasting lipids and prandial TGs | We will track this measure over a 5 week period. This may change as a patient's response to withdrawl and resumption of metformin varies

SECONDARY OUTCOMES:
• To provide a relative estimate of the composition of bile acids in bile sampled using the EnteroTest string | We will track this measure over a 5 week period. This may change as a patient's response to withdrawl and resumption of metformin varies
To measure sparse metformin profiles on the days when the PD endpoints are measured | We will track this measure over a 5 week period. This may change as a patient's response to withdrawl and resumption of metformin varies

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cambridge, Cambridgeshire, United Kingdom

REFERENCES:
- [Derived] Napolitano A, Miller S, Nicholls AW, Baker D, Van Horn S, Thomas E, Rajpal D, Spivak A, Brown JR, Nunez DJ. Novel gut-based pharmacology of metformin in patients with type 2 diabetes mellitus. PLoS One. 2014 Jul 2;9(7):e100778. doi: 10.1371/journal.pone.0100778. eCollection 2014. PMID 24988476
- See also: Results for study 114453 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/114453?search=study&search_terms=114453#rs